CLINICAL TRIAL: NCT03230591
Title: Impact of Agalsidase Alfa Therapy on Cardiac funcTION in Patients With Fabry's Cardiomyopathy (ACTION-Fabry Trial)
Brief Title: Impact of Agalsidase Alfa Therapy on Cardiac funcTION in Patients With Fabry's Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0471
Record Dates: First submitted 2017-07-21; First posted 2017-07-26 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Fabry Disease
Keywords: Fabry's disease; Agalsidase Alfa; Cardiomyopathy; Enzyme replacement therapy; Diastolic stress echocardiography; LV vortex flow; Cardiac MRI
MeSH Terms: conditions — Fabry Disease; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10cc blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry's disease: Fabry's disease patients who were confirmed by enzyme assay and gene study
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — LV vortex flow in Echocardiography

SUMMARY:
Study Design: This is an observational study. No treatment or intervention will be assigned to the subjects. All patients will receive full standard of care concomitant medication for the treatment of their cardiac condition. 25 patients with genetically confirmed Anderson-Fabry disease who have a plan to start ERT with Agalsidase Alfa will undergo 2D strain, diastolic stress echocardiography, LV vortex flow analysis, and CMR at baseline and after 1 year of treatment with ERT with Agalsidase Alfa for follow-up.

DETAILED DESCRIPTION:
1. Objectives - The purpose of this study is to evaluate the impact of ERT with Agalsidase Alfa on LV diastolic function and flow in patients with Fabry's cardiomyopathy using LV 2D strain, diastolic stress echocardiography, LV vortex flow and CMR.
2. Primary / Secondary Endpoint 1) Primary endpoint:

   * Change from baseline in peak exercise E/E' by diastolic stress echocardiography, global longitudinal strain and LV vortex flow parameters at 1 year 2) Secondary endpoints:
   * Changes from baseline in extracellular volume by CMR (T1 mapping) at 1 year follow up

     * Changes from baseline in evaluation of the degree of the resting LV diastolic function

       * Changes from baseline in other echo-parameters; LV mass index, reduction of peak exercise E/E prime at 1 year follow up

         * Changes from baseline in quality of life using questionnaire ⑤ Change from baseline in peak VO2, exercise time, AT by diastolic stress echocardiography at 1 year follow up ⑥ Change in T1 baseline (myo, ms) & T1 baseline (blood, ms), T1 postcontrast (myo, ms) & T1 baseline (blood, ms) by CMR
3. Study Methods 1) Study Design: This is an observational study. No treatment or intervention will be assigned to the subjects. All patients will receive full standard of care concomitant medication for the treatment of their cardiac condition. 25 patients with genetically confirmed Anderson-Fabry disease who have a plan to start ERT with Agalsidase Alfa will undergo 2D strain, diastolic stress echocardiography, LV vortex flow analysis, and CMR at baseline and after 1 year of treatment with ERT with Agalsidase Alfa for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16~ 75 years with Fabry disease confirmed by enzyme assay and gene test
* Patients who have LVH in 2D echocardiography (end diastolic septum and posterior wall thickness ≥ 12mm) or Patients who present with cardiac changes (indicative of disease progression such as decreased global longitudinal strain on 2D strain echocardiography or low native T1 mapping on CMR)
* Patients provided written informed consent to participate in this study

Exclusion Criteria:

* Contraindication for enzyme replacement treatment with Agalsidase Alfa
* Patients who cannot receive supine bicycle stress echocardiography, contrast echocardiography or CMR
* Patients with hemodynamically significant valvular heart disease or arrhythmias
* Patients who have history of acute myocardial infarction or congestive heart failure with reduced LV ejection fraction of less than 35%
* Patients who had any cerebrovascular accident in the prior 6 months
* Scheduled or planned surgery in the next 6 months
* Patients with chronic liver cirrhosis
* Patients who are allergic to contrast agent (e.g. Definity�, Lantheus Medical Imaging, North Billerica, MA, USA)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16 ~ 75 years with Fabry disease confirmed by enzyme assay and gene test
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
peak exercise E/E' by diastolic stress echocardiography | 1 year
  Change from baseline in peak exercise E/E' by diastolic stress echocardiography
global longitudinal strain | 1 year

SECONDARY OUTCOMES:
extracellular volume by CMR | 1 year
  Changes from baseline in extracellular volume by CMR (T1 mapping) at 1 year follow up
evaluation of the degree of the resting LV diastolic function | 1 year
  Changes from baseline in evaluation of the degree of the resting LV diastolic function
quality of life using questionnaire | 1 year
  Changes from baseline in quality of life using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided